CLINICAL TRIAL: NCT06862570
Title: Assessment of Local Anaesthesia Effectiveness Using Electric Pulp Tester in Symptomatic Irreversible Pulpitis Using 2% Lignocaine and 4% Articaine As Supplemental Anaesthetic Agents: an in Vivo Comparison
Brief Title: Assessment of Local Anaesthesia Effectiveness in Symptomatic Irreversible Pulpitis
Acronym: LA AGENTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 28 Military Dental Centre Lahore (Other Government)
Responsible Party: Principal Investigator, Zahra Zubair, Dr Zahra Zubair, 28 Military Dental Centre Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOCAL ANAESTHESIA
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Lignocaine, Articaine and Supplemental Buccal Infiltration
MeSH Terms: interventions — Lidocaine; Epinephrine; Carticaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2% LIGNOCAINE WITH EPINEPHRINE (Experimental): 1.8 ml of 2% Lignocaine with 1:100,000 epinephrine (36 mg/ml Lignocaine HCL, epinephrine bitartrate 0.0324 mg/ml)
  Interventions: Drug: 2% lignocaine with epinephrine 1.8 ml(36mg/ml lignocaine HCL, epinephrine bitartrate 0.0324mg/ml)
- 4% ARTICAINE WITH EPINEPHRINE (Experimental): 1.7 ml of 4% Articaine with 1:100,000 epinephrine (40mg/ml Articaine HCL, epinephrine bitartrate 0.018mg/ml)
  Interventions: Drug: 4% Articaine with epinephrine 1.7 ml (40mg/ml Articaine HCL, epinephrine bitartrate 0.018 mg/ml)

INTERVENTIONS:
Drug: 2% lignocaine with epinephrine 1.8 ml(36mg/ml lignocaine HCL, epinephrine bitartrate 0.0324mg/ml) — 2% lignocaine with epinephrine 1.8 ml(36mg/ml lignocaine HCL, epinephrine bitartrate 0.0324mg/ml)
  Other Names: HD caine Plus
  Arms: 2% LIGNOCAINE WITH EPINEPHRINE
Drug: 4% Articaine with epinephrine 1.7 ml (40mg/ml Articaine HCL, epinephrine bitartrate 0.018 mg/ml) — 4% Articaine with epinephrine 1.7 ml (40mg/ml Articaine HCL, epinephrine bitartrate 0.018 mg/ml)
  Other Names: Orabloc
  Arms: 4% ARTICAINE WITH EPINEPHRINE

SUMMARY:
This study aims to evaluate the comparative efficacy of two different local anaesthetic agents for supplemental buccal infiltration after a failed inferior alveolar nerve block in achieving profound pulpal anaesthesia for symptomatic irreversible pulpitis using 2% lignocaine and 4% articaine with vasoconstrictor epinephrine.

Alternate hypothesis:

There is a mean difference in local anaesthesia effectiveness of 2% lignocaine and 4% articaine containing epinephrine when used for buccal infiltration in pulpectomy of symptomatic irreversible pulpitis of mandibular posterior teeth after a failed inferior alveolar nerve block

DETAILED DESCRIPTION:
Patients diagnosed with symptomatic irreversible pulpitis are included in this study. Teeth will be divided into two groups after a failed inferior alveolar nerve block using 2% lignocaine containing 1:100,000 epinephrine. A sample size of 123, with the first group consisting of 62 patients, 2 cartridges of 32mg of 2% lignocaine with 1:100,000 epinephrine will be used for supplemental buccal infiltration. In group 2 of 61 patients, 40mg of 4% articaine with 1:100,000 epinephrine will be used. During the root canal treatment, a subjective assessment of lip anesthesia is recorded. An electric pulp tester is used for the evaluation of the presence or absence of pulpal anesthesia. A verbal analogue scale is also used to evaluate the presence or absence of pain.

After taking a brief history, informed consent will be taken. A rubber dam will be used. Electric pulp tester will be used on the control contralateral tooth, the experimental tooth preoperatively; after giving nerve block and achieving Lip numbness, the experimental tooth will again be evaluated with Electric pulp tester. An access cavity will be made. If there is still no pulpal anesthesia, supplemental anesthesia will be administered and Electric pulp tester will be used again.

A questionnaire containing a numerical rating scale will be given to each patient to record the intensity of pain felt after giving supplemental anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ages ranging from 18-to 55 years
2. Male/ Female
3. Mandibular posterior teeth with symptomatic irreversible pulpitis
4. Ability to understand the use of the pain scale
5. Patients with adequate oral hygiene and willing to participate in the study

Exclusion Criteria:

1. Any type of medication consumed before treatment
2. Patients who do not show profound lip numbness after giving inferior alveolar block
3. Periapical pathologies ( periapical abscess, sinus tract, periapical cyst, pulpal necrosis)
4. External resorption
5. Unfavorable location of the tooth, internal ankylosis, trismus, severe tooth malposition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Assessment of Local anaesthsia effectiveness in symptomatic irreversible pulpitis after afailed inferior alveolar nerve block using supplemental buccal infiltration | 5-10 minutes after administrating supplemental buccal infiltration
  Numeric Rating scale to assess absence or presence of pain after supplemental buccal infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Zubair, BDS, Principal Investigator — 28 Military Dental Centre
Locations (1):
- Zahra Zubir, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Gender, tooth no.
Time Frame: 6 months after publication
Access Criteria: zahra_zubair@hotmail.com

REFERENCES:
- [Background] Shapiro MR, McDonald NJ, Gardner RJ, Peters MC, Botero TM. Efficacy of Articaine versus Lidocaine in Supplemental Infiltration for Mandibular First versus Second Molars with Irreversible Pulpitis: A Prospective, Randomized, Double-blind Clinical Trial. J Endod. 2018 Apr;44(4):523-528. doi: 10.1016/j.joen.2017.10.003. Epub 2018 Feb 1. PMID 29397214
- [Background] Janiani P, Gurunathan D. Effectiveness of Pre-administered Natural Sweet-tasting Solution for Decreasing Pain Associated with Dental Injections in Children: A Split-mouth Randomized Controlled Trial. J Contemp Dent Pract. 2021 Dec 1;22(12):1434-1437. PMID 35656683
- [Background] Oghabi N, Renton T. Optimizing Local Anaesthetic Practice: Addressing Misconceptions and Minimizing Anaesthetic Failures. Dent Update. 2022;49(1):32-38.
- [Background] Martin E, Nimmo A, Lee A, Jennings E. Articaine in dentistry: an overview of the evidence and meta-analysis of the latest randomised controlled trials on articaine safety and efficacy compared to lidocaine for routine dental treatment. BDJ Open. 2021 Jul 17;7(1):27. doi: 10.1038/s41405-021-00082-5. PMID 34274944
- [Background] Dianat O, Mozayeni MA, Layeghnejad MK, Shojaeian S. The efficacy of supplemental intraseptal and buccal infiltration anesthesia in mandibular molars of patients with symptomatic irreversible pulpitis. Clin Oral Investig. 2020 Mar;24(3):1281-1286. doi: 10.1007/s00784-019-03006-8. Epub 2019 Jul 13. PMID 31302768
- [Background] Khan Q, Noor N, Anayat N, Khan TS, Ahmed M. Comparison Of Anaesthetic Efficacy Of Articaine And Lidocaine In Nonsurgical Endodontic Treatment Of Permanent Mandibular Molars With Symptomatic Irreversible Pulpitis. A Randomized Clinical Trial. J Ayub Med Coll Abbottabad. 2021 Apr-Jun;33(2):192-197. PMID 34137527